CLINICAL TRIAL: NCT06127953
Title: Intermediate Cleft Rhinoplasty in Unilateral Cleft Lip Patients: Approaches and Outcomes
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mohamed Elsayed Abdelmonem (Other)
Responsible Party: Sponsor-Investigator, Mohamed Elsayed Abdelmonem, Plastic surgery assistant lecturer, Sohag University
Organization: Sohag University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Soh-Med-23-10-09MD
Record Dates: First submitted 2023-11-04; First posted 2023-11-13 (Actual); Last update posted 2023-11-13 (Actual); Status verified 2023-11

CONDITIONS: Unilateral Cleft Lip
Keywords: Unilateral Cleft Lip; Cleft Rhinoplasty; Intermediate Cleft Rhinoplasty

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Unilateral Cleft Lip Patients (Other): Study is intermediate cleft rhinoplasty that will be performed in the patients with nasal deformities after repair of unilateral cleft lip congenital anomaly
  Interventions: Procedure: intermediate cleft rhinoplasty

INTERVENTIONS:
Procedure: intermediate cleft rhinoplasty — intermediate cleft rhinoplasty using open approach and combined techniques of Tajima, Dibbell and Potter's Rhinoplasty

SUMMARY:
This is a prospective study of 20 patients with unilateral cleft lip nasal deformity. The technique to be performed is open approach intermediate rhinoplasty using a hybrid technique combining Potter, Dibbell, and Tajima methods as needed (Potter 1954, Tajima and Maruyama 1977, Dibbell 1982). Lip revision will be performed with the intermediate cleft rhinoplasty according to the lip deformity if needed.

Aim of the work is To propose an algorithmic approach for management of unilateral cleft lip nasal deformity using hybrid techniques of intermediate cleft rhinoplasty and to assess the aesthetic and functional outcomes.

All the regulations of the ethical committee of the faculty of medicine in Sohag University will be followed. Each patient will have a private file with a non-disclosure policy at data presentation where all presented data do not contain any personal information specifying the identity of any of the patients. Informed written consent will be taken from all patients in the study.

Regarding patients' assessment, the following items will be fulfilled:

Full medical and operative history. Complete physical examination. Nasal examination, including nasal analysis, anterior rhinoscopy, Cottle maneuver, modified Cottle maneuver, and possibly endoscopic examination to fully assess any functional problems.

Routine laboratory investigations Standard preoperative photographs (frontal, lateral and basal).

Surgery follow up will be at 1 week ,1 month, 3 months, 6 months and 1 year and postoperative photographs will be taken.

DETAILED DESCRIPTION:
Cleft lip and palate is the most common congenital craniofacial abnormality (Jeong, Lee et al. 2012, Yue, Piao et al. 2023). Cleft nasal deformity is the most prominent aesthetic problem in the growing cleft patient after lip repair (Park, Koo et al. 2022). Correction of the residual cleft lip nasal deformity remains a complex and difficult to manage challenge as nasal asymmetry increases with the growth and development of the affected child in addition to the scarring from previous surgeries of the lip and nose (Ayeroff, Volpicelli et al. 2019). The cleft nasal deformity affects all layers of the nose including the bony platform, the inner lining, the cartilaginous infrastructure, and the external skin (Olds and Sykes 2022). The severity of nasal deformity is dependent upon the degree of the original cleft lip abnormality (Gary and Sykes 2016).

There has been a debate for long time regarding the timing of cleft rhinoplasty and there has been a trend to perform it after the age of full maturity. The rationale behind this belief was to avoid interference with nasal growth, however many studies have disproved this traditional idea (Pagan, Sterling et al. 2021) and even in Millard's classic paper, he pointed out that a minor aesthetic correction during childhood is sometimes required (Millard 1964). Cleft rhinoplasties are divided into 3 stages: primary, performed within the first year of life; intermediate, performed prior to completion of facial growth; and definitive, which occurs after skeletal and dental maturity (Ayeroff, Volpicelli et al. 2019).

Intermediate cleft rhinoplasty is defined as any nasal surgery performed between the time of initial cleft lip repair and the time at which the patient reaches facial skeletal maturity (around 15 to 17 years of age in females and in male patients at approximately 16 to 18 years of age) (Gary and Sykes 2016). Intermediate rhinoplasty is indicated in case of functional compromise (nasal obstruction and sleep apnea) as in severe septal deviation and severe alar deformities and in situations of child and parent wishes due to psychological distress from their peers in school age. Some studies have shown that children with orofacial cleft suffer the highest incidence of depression, anxiety, and negative peer relationships around the ages 8 to 10 years (Hoshal, Solis et al. 2020, Olds and Sykes 2022, Park, Koo et al. 2022).

One of the earliest attempts to correct the nasal tip deformity was in 1932 when Gillies and Kilner described the "alar shift" technique, allowing for the advancement of the cleft side columella towards the tip (Wilkie 1969). In 1938, McIndoe was the first surgeon to reposition and fix the cartilage of the cleft side (McIndoe 1938), but Potter in 1954 added the concept of not only repositioning the lower lateral cartilage medially but also the lateral release via an open nasal approach(Potter 1954, Rousso 2015).

In 1964, Millard introduced the concept of additional support using auricular cartilage grafts at 5 years of age with cleft tip revisions (Millard 1964). Tajima and Maruyama in 1977 pointed out that the overhanging alar web is one of the most visible stigmata of cleft noses and this excess skin will result in cartilage malposition and redundancy (Tajima and Maruyama 1977, Nicksic, Pfaff et al. 2018). In 1982, Dibbell described a procedure to address the alar web by rotating and advancing the nostril medially and superiorly in addition to fixation of cleft lower lateral cartilage (Dibbell 1982). Blackwell in 1985 focused on both cartilage reposition and utility of additional support (Blackwell, Parry et al. 1985, Nicksic, Pfaff et al. 2018).

Cutting in 2009 described a technique for tip cleft rhinoplasty which combines an open rhinoplasty with the Dibbell and Tajima techniques (Flores, Sailon et al. 2009). Ayeroff, Volpicelli et al. described the component restoration approach for intermediate cleft rhinoplasty that addresses the three anatomical disturbances of the cleft nasal tip: lower lateral cartilage malpositioning, lower lateral cartilage hypoplasia, and nasal lining deficiency(Ayeroff, Volpicelli et al. 2019). Ohara, Nakajima et al. described the use of the subcutaneous flap technique to address the cleft bulbous nasal tip and define the alar groove through an open rhinoplasty approach (Ohara, Nakajima et al. 2009).

There are conflicting views regarding the use of cartilage grafts in intermediate cleft rhinoplasty. However, recent studies approved their use during the 5- to 13-year age period and found that it was effective in aesthetic and functional outcomes, with a low-risk profile (Ozaki, Chaffoo et al. 2006, Lu, Yao et al. 2017, Zhang, Bai et al. 2018, Pagan, Sterling et al. 2021).

The large number of techniques in the literature to address this challenge is a testament to both the complexity of the task and the limitations of our ability to provide dependable surgical solutions (Hoshal, Solis et al. 2020). Successful surgical correction is often surgeon-dependent and often based on training and experience (Hoshal, Solis et al. 2020). As Dibbell observed in 1982, "Anytime there are many differing attacks on a surgical problem area, the sophisticated practitioner will conclude that none of these approaches are satisfactory" (Dibbell 1982). To date, there is no consensus regarding universal guidelines or the ideal techniques for the management of cleft nasal deformities (Olds and Sykes 2022).

ELIGIBILITY:
Inclusion Criteria:

* Patients with repaired unilateral cleft lip with or without cleft palate with residual nasal deformity.
* Patients aged 1 to 13 years.
* Patients who underwent or did not undergo primary rhinoplasty during the cleft lip repair.

Exclusion Criteria:

* Patients with bilateral cleft lip.
* Patients who underwent lip/nose revision.
* Patients or parents' refusal to participate in the study.

Ages: 1 Year to 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Estimated)
Dates: Start 2023-10-23 (Actual); Primary Completion 2024-10-23 (Estimated); Study Completion 2025-01-23 (Estimated)

PRIMARY OUTCOMES:
measurements of nostril apex height on the cleft lip side. | 1 week then 1, 3, 6 and 12 months post operative date
  Preoperative and postoperative measurements of nostril apex height on the cleft lip side will be compared to determine the effects of surgery on the nasal form.

SECONDARY OUTCOMES:
The visual effect of the rhinoplasty. | 1 week then 1, 3, 6 and 12 months post operative date
  The visual effect of the operation will also be assessed according to the Global Aesthetic Improvement Scale (GAIS) which is a simple five-point scale to be determined by the patient or patient's parents for assessing global aesthetic improvement in appearance of the nose compared to pretreatment. The five points are: "1" is very much improved, "2" is much improved, "3" is improved, "4" is no change and "5" is worse.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Medicine Sohag University, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ayeroff JR, Volpicelli EJ, Mandelbaum RS, Pfaff MJ, Asanad S, Bradley JP, Lee JC. Component Restoration in the Unilateral Intermediate Cleft Tip Rhinoplasty: Technique and Long-Term Outcomes. Plast Reconstr Surg. 2019 Mar;143(3):572e-580e. doi: 10.1097/PRS.0000000000005367. PMID 30601327
- [Background] Gary C, Sykes JM. Intermediate and Definitive Cleft Rhinoplasty. Facial Plast Surg Clin North Am. 2016 Nov;24(4):487-494. doi: 10.1016/j.fsc.2016.06.017. PMID 27712816
- [Background] Hoshal SG, Solis RN, Tollefson TT. Controversies in Cleft Rhinoplasty. Facial Plast Surg. 2020 Feb;36(1):102-111. doi: 10.1055/s-0040-1701477. Epub 2020 Mar 19. PMID 32191966
- [Background] Blackwell SJ, Parry SW, Roberg BC, Huang TT. Onlay cartilage graft of the alar lateral crus for cleft lip nasal deformities. Plast Reconstr Surg. 1985 Sep;76(3):395-401. doi: 10.1097/00006534-198509000-00010. PMID 4034756
- [Background] Nicksic PJ, Pfaff MJ, Ayeroff JR, Lee JC. Management of the Cleft Nasal Tip: An Overview of Classic Techniques and Strategies. Ann Plast Surg. 2018 May;80(5):581-586. doi: 10.1097/SAP.0000000000001334. PMID 29389706